CLINICAL TRIAL: NCT03435328
Title: Hyposalivation Response To Transcutaneous Electrical Nerve Stimulation In Diabetic Type 2 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/001504
Record Dates: First submitted 2018-01-27; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Diabetes type2; Hyposalivation
Keywords: TENS
MeSH Terms: conditions — Xerostomia | interventions — Transcutaneous Electric Nerve Stimulation

ARMS (1):
- TENS intervention (Experimental): one group receiving TENS:
  - The electrode of TENS unit will be placed vertically, externally on skin overlying the parotid gland, in the preauricular area bilaterally, 1 cm in front of the tragus area.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — * Duration of stimulation: 5 minutes.
  * Frequency: will be fixed at 50 Hertz.
  * Pulse duration: 250 µs.
  * Intensity: optimal intensity of TENS (amplitude will be gradually increased to the maximum intensity that the subject will be comfortable and tolerate it).
  * Sessions: only one session

SUMMARY:
This study evaluates response of abnormal low salivary flow rate to transcutaneous electrical nerve stimulation (TENS) in diabetic type 2 patients. Response of saliva monitored for all participants receiving only one session of 5-minute extraoral TENS on bilateral parotid glands.

DETAILED DESCRIPTION:
Diabetes mellitus is the most significant disorder associated with varied oral manifestation ranging from xerostomia (subjective sensation od dry mouth) to serious bacterial and fungal infections due to alterations in flow rate of saliva.

Systemic agents increase rate of stimulated salivary flow but often have unfavourable side effects such as profuse sweating, rhinitis, dyspepsia.

Use of TENS in stimulation of saliva has been studied in the past which showed moderate promising results. However, it never became a part of the mainstream therapy of hyposalivation.

It has been postulated that transcutaneous electric nerve stimulation (TENS) could directly stimulate the auriculotemporal nerve, which supplies the parotid gland, whereas it remains unclear whether there is also an indirect action (via afferent pathways) onto the salivary reflex arch.

Starting a prevention program as early as possible considering the most practical, cost effective and efficient treatments with the best risk-benefit ratio will help to diminish dry mouth symptoms and sequelae (intraoral and extraoral complications).

ELIGIBILITY:
Inclusion Criteria:

1. non-smoker diabetic patients type II
2. Patients with unstimulated resting saliva ≤ 0.16 ml/min considered to be abnormally low flow rate and included in the study (Navazesh et al., 1992)

Exclusion Criteria:

* Cancer patients (patients on chemotherapy/immunotherapy and history of head and neck radiotherapy).
* Cardiac patients (cardiac pacemakers and defibrillators).
* Patients wearing hearing aids.
* Chronic inflammatory autoimmune diseases
* Acute oral inflammatory disorders
* Patients with neurological disorders.
* Habits (mouth breathing, smoking, alcohol and drug abuse).
* Salivary gland diseases and disorders.
* Psychogenic diseases.
* Endocrine diseases.
* Patients undergoing pharmacological management for xerostomia.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
salivary volume | After only one session of five-minutes TENS
  It is estimated as follow:
  * The patients advised to have nothing to eat, drink, chew gum, intake coffee and oral hygiene before the test.
  * whole resting salivary volume (ml) planned to be performed using low forced spitting technique in graduated test tube before TENS application.
  * stimulated salivary volume (ml) collected after TENS application is compared to whole resting salivary volume to assess improvement. .

SECONDARY OUTCOMES:
salivary flow rate | After only one session of five-minutes TENS
  It is estimated as follow:
  * By dividing whole resting salivary volume on five minute collection period , thus whole resting salivary flow rate (ml/minute) is obtained.
  * Dividing stimulated salivary volume - collected after TENS application - on five minute collection period, thus stimulated salivary flow rate (ml/minute) is obtained.
  * Assessing improvement is done by comparing stimulated with whole resting salivary flow rate.
Eight-item visual analogue scale xerostomia questionnaire | After only one session of five-minutes TENS
  * Visual analogue scale is a horizontal line,100 millimeters (mm) in length and anchored by word descriptors at each end.
  * Items are "Rate the difficulty you experience in swallowing due to dryness", "Rate the difficulty you experience in speaking due to dryness","Rate how much saliva is in your mouth","Rate the dryness of your mouth", "Rate the dryness of your throat", "Rate the dryness of your lips", "Rate the dryness of your tongue" ," Rate the level of your thirst" respectively.
  * Before and after treatment, the researcher ask each item to the patient.Then, the patient ts asked to mark his response (perception of his current state) for the item by placing a vertical line on the scale of each item.
  * The researcher determine scale score response of each item by measuring distance in mm.
  * Decreased post-treatment of visual analogue scale score for each item considered improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Hala MH Ezz-eldeen, Professor, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No